CLINICAL TRIAL: NCT07017140
Title: Immersive Functional Virtual Reality in People With Acquired Brain Injury and Unilateral Spatial Neglect: A Feasibility and Usability Study
Brief Title: Immersive Functional Virtual Reality in People With Acquired Brain Injury and Unilateral Spatial Neglect
Acronym: REVINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Hospital Vall d'Hebron (Other); Consorci Hospitalari de Vic (CHV) (Unknown)
Responsible Party: Principal Investigator, Josan Merchan, Dr. Josan Merchan-Baeza, University of Vic - Central University of Catalonia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25/009
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Acquired Brain Injury Including Stroke; Unilateral Spatial Neglect (USN); Stroke; Traumatic Brain Injury
Keywords: acquired brain injury; unilateral spatial neglect; stroke; traumatic brain injury; cognitive and motor rehabilitation; virtual reality-based therapy; virtual reality
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm feasibility study using a single-group interrupted time series design. All participants receive the same intervention: 12 sessions of immersive functional virtual reality (IFVR) over 4 weeks. Pre- and post-intervention outcomes are assessed at three time points each, spaced one month apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 - Immersive Functional Virtual Reality (Experimental): Participants will receive 12 individual IFVR sessions (30 minutes each, 3 sessions per week for 4 weeks) using the KINESIX system. The intervention targets visuospatial attention and upper limb function through progressive, gamified exercises in a controlled virtual environment. Sessions are supervised by a physiotherapist or occupational therapist. In addition to the VR intervention, participants continue their usual care rehabilitation as prescribed at their center.
  Interventions: Device: Immersive Functional Virtual Reality Intervention using a Head-Mounted Display System for Spatial Neglect Rehabilitation

INTERVENTIONS:
Device: Immersive Functional Virtual Reality Intervention using a Head-Mounted Display System for Spatial Neglect Rehabilitation — Participants receive 12 sessions (30 minutes each, 3 per week over 4 weeks) of immersive functional virtual reality (IFVR) using the KINESIX system, a CE-certified Class I head-mounted display device. The intervention targets visuospatial attention and upper limb function through progressively challenging, gamified exercises. All sessions are supervised by a physiotherapist or occupational therapist and delivered in a safe, controlled rehabilitation setting. Participants continue receiving usual care.

SUMMARY:
Unilateral spatial neglect (USN) is a common and highly disabling condition following acquired brain injury (ABI), significantly impairing individuals' ability to perform daily activities and reducing their autonomy. It frequently affects patients who have suffered a stroke or traumatic brain injury, and it is often associated with worse functional outcomes and increased care needs. Despite advances in neurorehabilitation, conventional assessment and treatment tools for USN have shown limitations in sensitivity and ecological validity.

Immersive Functional Virtual Reality (IFVR) is an emerging and promising technology that creates controlled, interactive environments, facilitating both assessment and rehabilitation in a motivating and safe way. The REVINE study explores the feasibility, usability, and preliminary clinical effects of an immersive VR-based intervention tailored to address motor and spatial deficits in adults with ABI and USN.

This is a prospective, non-controlled feasibility study using a single-group interrupted time series design. Participants (N=30) will be recruited from two neurorehabilitation services in Catalonia (Spain): the Neurological Rehabilitation and Brain Injury Unit at Vall d'Hebron University Hospital and the Outpatient Rehabilitation Service at Consorci Hospitalari de Vic. Eligible participants will be adults with ABI in the subacute or chronic phase, presenting USN (as measured by the Catherine Bergego Scale and the Bells Cancellation Test) and mild-to-moderate upper limb impairment.

The intervention consists of 12 supervised individual IFVR sessions (30 minutes/session, 3 times/week for 4 weeks), using the KINESIX system (NeuroGroup XR Inc., Montreal, Canada). A progressive series of gamified tasks will be delivered through immersive VR, targeting spatial exploration and upper limb function, with adjustable difficulty and real-time feedback.

Participants will undergo three pre-intervention and three post-intervention evaluations, spaced one month apart. Clinical outcomes include the degree of USN (measured by the Catherine Bergego Scale, the Bells Cancellation Test, and the KINESIX light-reaching test), usability (System Usability Scale), and satisfaction (User Satisfaction Evaluation Questionnaire). Feasibility outcomes include recruitment and retention rates, adherence to treatment, session completion times, adverse events, and therapist assistance level.

We hypothesize that IFVR will be a viable and well-accepted intervention, with high user satisfaction, minimal adverse effects, and measurable improvements in neglect-related outcomes. This study aims to inform the future design of larger-scale trials and support the integration of IFVR into routine neurorehabilitation settings or home-based telerehabilitation programs.

DETAILED DESCRIPTION:
Background and Rationale

Acquired brain injury (ABI), including stroke and traumatic brain injury, is a leading cause of long-term disability worldwide. One of its most disabling consequences is unilateral spatial neglect (USN), a complex perceptual-attentional syndrome characterized by an impaired ability to attend, respond, or orient to stimuli presented on the side opposite the brain lesion. USN significantly affects functional independence and daily living activities such as grooming, eating, dressing, or mobility, and it is associated with a poorer rehabilitation prognosis and prolonged dependence on caregivers.

Despite the high prevalence and impact of USN, conventional assessment tools (e.g., cancellation tasks, line bisection) often lack sensitivity to detect subtle deficits and do not reflect real-life performance. Furthermore, traditional rehabilitation approaches may be insufficient to address the multifaceted nature of USN, especially its extrapersonal and representational aspects.

Virtual reality (VR) technologies provide controlled, interactive environments that simulate real-life situations, enabling both the assessment and treatment of cognitive and motor impairments. Immersive Functional Virtual Reality (IFVR), in particular, can engage users in multisensory, gamified tasks that promote neuroplasticity while ensuring ecological validity. Previous evidence supports the use of VR-especially semi-immersive systems-for USN rehabilitation, though immersive systems remain underexplored in clinical trials and feasibility studies.

Study Objectives

The REVINE project aims to evaluate the feasibility, usability, and preliminary clinical effects of an IFVR intervention in adults with ABI and USN.

The general objectives of the REVINE project are:

* GO1. To describe the feasibility of using immersive functional virtual reality (IFVR) for the rehabilitation of individuals with unilateral spatial neglect (USN) following acquired brain injury (ABI).
* GO2. To describe the usability of IFVR among individuals with USN after ABI.
* GO3. To evaluate the applicability of IFVR as an assessment tool for USN in individuals with ABI.
* GO4. To assess the clinical effects of IFVR on USN in people with ABI.

The specific objectives are:

* SO1. To describe recruitment and consent rates, as well as participant retention throughout the study.
* SO2. To record treatment adherence based on the number of sessions attended versus those planned.
* SO3. To quantify the time spent during intervention and assessment sessions.
* SO4. To record the type, severity, and duration of potential adverse events during treatment.
* SO5. To document the time spent according to the type of game used and its level of difficulty.
* SO6. To analyse the level of therapist assistance required during intervention sessions.
* SO7. To determine perceived usability using the System Usability Scale (SUS).
* SO8. To describe user satisfaction with the IFVR intervention using the User Satisfaction Evaluation Questionnaire (USEQ).
* SO9. To evaluate the clinical effect of IFVR on USN severity using the Bells Cancellation test, the Catherine Bergego Scale (CBS), and the KINESIX light test.

Study Design

This is a prospective, single-arm feasibility study employing a single interrupted time series design. A total of 30 participants will be recruited using a non-probabilistic convenience sampling method. Each participant will undergo three pre-intervention evaluations (T1, T2, T3) and three post-intervention evaluations (T4, T5, T6), each spaced one month apart. The intervention will consist of 12 individual, supervised IFVR sessions over four weeks (three sessions per week, 30 minutes per session).

Setting and Participants

The study will take place at two specialized rehabilitation centers in Catalonia, Spain:

* The Neurological Rehabilitation and Brain Injury Unit at Vall d'Hebron University Hospital (Barcelona).
* The Outpatient Rehabilitation Service of the Consorci Hospitalari de Vic (Vic, Barcelona).

Eligible participants must meet the following criteria:

* Adults (≥18 years) with a diagnosis of ABI in the subacute (>7 days to 6 months) or chronic phase (>6 months).
* Presence of USN (≥6 omissions in the Bells Cancellation Test).
* Mild to moderate upper limb impairment (Fugl-Meyer Upper Extremity >29).
* Medically stable and capable of participating in rehabilitation.

Exclusion criteria include severe cognitive, visual, or auditory deficits, language comprehension difficulties, hypersensitivity or intolerance to VR headsets, photosensitive epilepsy, or active behavioral disturbances.

Intervention

The IFVR intervention will be delivered using the KINESIX system (NeuroGroup XR Inc.), consisting of a VR headset with integrated software, a therapist tablet interface, and a web-based monitoring platform. The intervention includes 12 exercises grouped into three modules: practice, activities, and participation. Tasks will focus on visuospatial exploration, reaching, grasping, and manipulating virtual objects, particularly in the contralesional space.

Exercises are designed with five increasing difficulty levels to support motor learning and maintain user engagement. Playlists of exercises will progress in difficulty as the participant advances through sessions. Sessions will take place in a safe space under the supervision of a physiotherapist or occupational therapist.

Outcome Measures

Feasibility Outcomes:

* Recruitment, consent, and retention rates.
* Session adherence and duration.
* Frequency and severity of adverse events.
* Level of therapist assistance (7-point Likert scale).

Usability and Satisfaction:

* System Usability Scale (SUS): 10-item Likert scale, score range 0-100.
* User Satisfaction Evaluation Questionnaire (USEQ): 6-item Likert scale, average score 1-7.

Clinical Outcomes:

* Catherine Bergego Scale (CBS): Assesses functional neglect in daily activities (score 0-30).
* Bells Cancellation Test: Screening tool for visual neglect (≥6 omissions indicates USN).
* KINESIX Light Reach Test: Measures spatial reach using 209 LED lights to assess peripersonal and extrapersonal attention.

Safety Considerations

Initial familiarization with the VR headset will ensure gradual exposure to immersive environments. Any adverse events (e.g., dizziness, nausea) will be documented and managed using a pre-defined protocol. Sessions may be interrupted or modified based on participant tolerance. All devices will be disinfected between uses.

Timeline

The study will span 24 months, starting in December 2024. Recruitment will begin in March 2025, following ethics approval, and continue for approximately 12 months. Post-intervention follow-up will conclude by late 2026. Data analysis is planned for November 2026 to January 2027.

Significance and Innovation

This study will provide essential insights into the practical implementation of immersive VR technologies in neurorehabilitation settings. By focusing on feasibility and user experience, the REVINE project seeks to bridge the gap between experimental innovation and clinical application. The findings will inform the design of future randomized controlled trials and the potential integration of IFVR into conventional and remote rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosis of acquired brain injury (stroke or traumatic brain injury) in the subacute phase (>7 days to 6 months) or chronic phase (>6 months).
* Presence of unilateral spatial neglect, defined as omission of 6 or more bells on the left hemifield in the Bells Cancellation Test.
* Currently receiving care at the Outpatient Rehabilitation Service of the Consorci Hospitalari de Vic or at Vall d'Hebron University Hospital, or listed in the historical patient registry of these centers.
* Presence of mild to moderate upper limb impairment, defined as a score >29 on the Fugl-Meyer Upper-Extremity scale.
* Medically stable and eligible to begin a rehabilitation program.
* Willing to participate in the study and able to provide signed informed consent.

Exclusion Criteria:

* Delirium and/or behavioral disturbances that prevent the participant from following simple instructions.
* Severe cognitive impairment, defined as a Mini-Mental State Examination (MMSE) score below 18, that interferes with the use of virtual reality.
* Severe visual and/or auditory impairment that prevents the use of immersive VR goggles.
* Severe language comprehension difficulties that interfere with the instructions during the intervention.
* Hypersensitivity that prevents the placement of the VR headset.
* Headache or dizziness induced by the use of VR goggles.
* History of photosensitive epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the immersive virtual reality intervention | From enrollment to T6 (final follow-up, 5 months after baseline)
  Feasibility will be assessed based on:
  * Recruitment rate: number of participants enrolled versus eligible.
  * Consent rate: number of participants agreeing to participate after invitation.
  * Retention rate: percentage completing all planned assessments.
  * Adherence: number and percentage of VR sessions completed out of 12.
  * Adverse events: type, severity, and frequency of VR-related events.
  * Therapist assistance level: rated on a 7-point Likert scale from full dependence to full independence.

SECONDARY OUTCOMES:
System Usability (System Usability Scale - SUS) | At T4 (first post-intervention evaluation, 3 months after baseline)
  Usability of the immersive virtual reality system will be evaluated using the System Usability Scale (SUS), a 10-item questionnaire scored on a 0-100 scale. Scores above 68 indicate acceptable usability.
User Satisfaction (User Satisfaction Evaluation Questionnaire - USEQ) | At T4 (first post-intervention evaluation, 3 months after baseline)
  Participant satisfaction with the intervention will be assessed using the USEQ, a 6-item scale rated on a 7-point Likert scale. Scores range from 1 (low satisfaction) to 7 (high satisfaction).
Change in Unilateral Spatial Neglect (Catherine Bergego Scale) | From T1 (baseline) to T6 (first post-intervention evaluation, 5 months after baseline)
  Spatial neglect will be assessed using the Catherine Bergego Scale (CBS), a 10-item observational scale that evaluates the impact of neglect on daily activities. Each item is scored from 0 (no neglect) to 3 (severe neglect); total scores range from 0 to 30, with higher scores indicating more severe neglect.
Change in Unilateral Spatial Neglect (Bells Cancellation Test) | From T1 (baseline) to T6 (first post-intervention evaluation, 5 months after baseline)
  The Bells Cancellation Test measures visual neglect by asking participants to identify 35 bell figures among distractors on a structured sheet. Omission of 6 or more bells on the left side suggests unilateral spatial neglect. The total number and spatial distribution of omissions will be recorded and compared between time points.
Change in Spatial Reach (KINESIX Light Reach Test) | From T1 (baseline) to T6 (first post-intervention evaluation, 5 months after baseline)
  Spatial reach and exploration will be measured using the KINESIX Light Reach Test, a VR-based assessment involving activation of LED lights on a horizontal surface. The number and location of lights reached will be recorded to evaluate performance in peripersonal and extrapersonal space.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jose Antonio Merchan-Baeza, PhD, Principal Investigator — University of Vic - Central University of Catalonia
Locations (2):
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona, Spain
  - Consorci Hospitalari de Vic, Vic, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the exploratory nature of this feasibility study and the limited sample size. Additionally, the study involves sensitive health data from individuals with acquired brain injury, and the data use has been approved only for internal analysis within the research team under strict confidentiality agreements. No extended consent for data sharing beyond the current project scope has been obtained.

REFERENCES:
- [Background] Hategeka C, Ruton H, Karamouzian M, Lynd LD, Law MR. Use of interrupted time series methods in the evaluation of health system quality improvement interventions: a methodological systematic review. BMJ Glob Health. 2020 Oct;5(10):e003567. doi: 10.1136/bmjgh-2020-003567. PMID 33055094
- [Background] Gammeri R, Iacono C, Ricci R, Salatino A. Unilateral Spatial Neglect After Stroke: Current Insights. Neuropsychiatr Dis Treat. 2020 Jan 10;16:131-152. doi: 10.2147/NDT.S171461. eCollection 2020. PMID 32021206
- [Background] Corbetta M, Kincade MJ, Lewis C, Snyder AZ, Sapir A. Neural basis and recovery of spatial attention deficits in spatial neglect. Nat Neurosci. 2005 Nov;8(11):1603-10. doi: 10.1038/nn1574. Epub 2005 Oct 23. PMID 16234807
- [Background] Cavedoni S, Cipresso P, Mancuso V, Bruni F, Pedroli E. Virtual reality for the assessment and rehabilitation of neglect: where are we now? A 6-year review update. Virtual Real. 2022;26(4):1663-1704. doi: 10.1007/s10055-022-00648-0. Epub 2022 May 30. PMID 35669614
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed Definitions and a Shared Vision for New Standards in Stroke Recovery Research: The Stroke Recovery and Rehabilitation Roundtable Taskforce. Neurorehabil Neural Repair. 2017 Sep;31(9):793-799. doi: 10.1177/1545968317732668. PMID 28934920